CLINICAL TRIAL: NCT01678079
Title: Bioavailability and Acceptability of Enteric-Coated Microencapsulated Calcium During Pregnancy: A Randomized Crossover Trial in Bangladesh (Encapsulated Calcium Absorption in Pregnancy)
Brief Title: Encapsulated Calcium Absorption in Pregnancy
Acronym: ENCAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Baylor College of Medicine (Other); Johns Hopkins Bloomberg School of Public Health (Other); Saving Lives at Birth (Unknown); Grand Challenges Canada (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); Government of Norway (Unknown); Bill and Melinda Gates Foundation (Other); World Bank (Other)
Responsible Party: Principal Investigator, Daniel Roth, Staff Physician, Paediatric Medicine, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1000033463
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Pregnancy
Keywords: Pregnancy; Micronutrient Powder; Calcium; Iron; Bangladesh

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Micronutrient Powder, Enteric-coated Calcium (500 mg/day) (Experimental): Encapsulated Calcium
  Interventions: Dietary Supplement: Encapsulated Calcium
- Micronutrient Powder, Enteric-coated Calcium (1000 mg/day) (Experimental): Encapsulated Calcium
  Interventions: Dietary Supplement: Encapsulated Calcium
- Micronutrient Powder, Enteric-coated Calcium (1500 mg/day) (Experimental): Encapsulated Calcium
  Interventions: Dietary Supplement: Encapsulated Calcium
- Micronutrient Powder, Uncoated Calcium (500 mg/day) (Active Comparator): Non-capsulated Calcium
  Interventions: Dietary Supplement: Non-capsulated Calcium
- Micronutrient Powder, Uncoated Calcium (1000 mg/day) (Active Comparator): Non-capsulated Calcium
  Interventions: Dietary Supplement: Non-capsulated Calcium
- Micronutrient Powder, Uncoated Calcium (1500 mg/day) (Active Comparator): Non-capsulated Calcium
  Interventions: Dietary Supplement: Non-capsulated Calcium

INTERVENTIONS:
Dietary Supplement: Encapsulated Calcium — The intervention is a multi-micronutrient powder containing enteric-coated calcium carbonate, in addition to ferrous fumarate (60 mg of elemental iron) and folic acid (400 µg).
  Arms: Micronutrient Powder, Enteric-coated Calcium (1000 mg/day); Micronutrient Powder, Enteric-coated Calcium (1500 mg/day); Micronutrient Powder, Enteric-coated Calcium (500 mg/day)
Dietary Supplement: Non-capsulated Calcium — The comparator/control intervention is a micronutrient powder containing non-coated calcium (500, 1000 or 1500 mg elemental calcium from calcium carbonate), ferrous fumarate (60 mg of elemental iron) and folic acid (400 µg). This product will be similar in Ca dose, appearance, taste and texture to the experimental formulation but will not include the enteric-coating.
  Arms: Micronutrient Powder, Uncoated Calcium (1000 mg/day); Micronutrient Powder, Uncoated Calcium (1500 mg/day); Micronutrient Powder, Uncoated Calcium (500 mg/day)

SUMMARY:
This study will enroll at least 60 pregnant women in a randomized cross-over study in Dhaka, Bangladesh. Each participant will be randomized to one of 3 calcium doses: 500 mg, 1000 mg, 1500 mg elemental Ca per day. Each participant will undergo two calcium absorption tests, one with a micronutrient supplement powder containing non-encapsulated (non-coated) calcium and the other with a micronutrient supplement powder containing encapsulated calcium at the same dose. The absorption tests will be separated by a 2-week washout period. Fractional calcium absorption will be measured using the dual stable isotope method. For each test, the formulation will be administered orally for 9 days; on the 10th day, a 44Ca- labeled stable isotope will be given orally and a 42Ca-labeled stable isotope dose will be given intravenously. Urine will be collected for 48 hours to measure calcium absorption.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 30 years
* Current residence in Dhaka at a fixed address
* Plan to remain in Dhaka for at least 2 months from date of enrolment
* Gestational age of 27 completed weeks ± 1 week, estimated based on the recalled first day of the last menstrual period (LMP)

Exclusion Criteria:

* Complicated medical or obstetric history, based on self-report or clinical assessment by physician (e.g., cardiovascular disease, uterine hemorrhage, placenta previa, threatened abortion, hypertension, preeclampsia, multiple gestation, diabetes, renal disease)
* Higher risk pregnancy based on one or more of the following clinical findings at time of recruitment:

  * Severe anemia (hemoglobin <70 g/L assessed by Hemocue)
  * Proteinuria (≥ 100 mg/dl based on urine dipstick)
  * Glycosuria (≥ 100 mg/dl based on urine dipstick)
  * Hypertension (systolic blood pressure, ≥140 mm Hg and/or diastolic blood pressure ≥90 mm Hg)
* Reported use of dietary supplements that contain >500 mg of calcium per day and/or >400 IU (10 mcg) of vitamin D per day
* Reported use (chewing) of betel leaf, areca nut and lime (together referred to locally as paan) during pregnancy

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Fractional Calcium Absorption | Fractional calcium absorption during day 10-11
  The primary analysis will be a comparison of mean fractional absorption of the two calcium formulations (enteric-coated vs. non-coated). The secondary analysis will be a comparison of mean fractional absorption across different calcium doses (500, 1000, 1500 mg per day).
Fractional Calcium Absorption | Fractional calcium absorption during day 35-36
  The primary analysis will be a comparison of mean fractional absorption of the two calcium formulations (enteric-coated vs. non-coated). The secondary analysis will be a comparison of mean fractional absorption across different calcium doses (500, 1000, 1500 mg per day).

SECONDARY OUTCOMES:
Palatability and Acceptability | Baseline, +10/11 days, +35/36 days
  The palatability and acceptability of the microencapsulated and non-encapsulated calcium formulations will be surveyed to assess the following parameters using semi-quantitative measures (i.e. Organoleptic properties, such as taste, odour, texture and colour, and adherence to prescribed micronutrient regimen, and reasons for non-adherence)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roth, MD, Principal Investigator — The Hospital for Sick Children; Stanley Zlotkin, MD, Principal Investigator — The Hospital for Sick Children
Locations (4):
- United States (2):
  - The Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - Baylor College of Medicine, Houston, Texas
- International Center for Diarrheal Disease Research, Dhaka, Bangladesh
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Roth DE, Pezzack B, Al Mahmud A, Abrams SA, Islam M, Aimone Phillips A, Baxter JA, Dimitris MC, Hawthorne KM, Ahmed T, Zlotkin SH. Bioavailability of enteric-coated microencapsulated calcium during pregnancy: a randomized crossover trial in Bangladesh. Am J Clin Nutr. 2014 Dec;100(6):1587-95. doi: 10.3945/ajcn.114.090621. Epub 2014 Oct 1. PMID 25411294